CLINICAL TRIAL: NCT03260686
Title: The Effectiveness of Video Guided Exercise After Stroke
Brief Title: Video Guided Exercise After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Carl Thompson, Professor Carl Thompson, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT16/188(HRA)
Record Dates: First submitted 2017-08-18; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cerebral Stroke ,Cerebrovascular Accident, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Video Guided Group (Experimental): Participants receive standard care physiotherapy for their upper limb rehabilitation, with exercises given either verbally or in writing as decided by the prescribing clinician. In addition the participants will receive a personalised video guide of their exercises, filmed during their therapy session to use for independent practice when back on the ward.
  Interventions: Other: experimental
- Treatment as usual (No Intervention): Participants receive standard care physiotherapy for their upper limb rehabilitation, with exercises given either verbally or in writing as decided by the prescribing clinician

INTERVENTIONS:
Other: experimental — video guide for upper limb exercise
  Arms: Video Guided Group

SUMMARY:
People who have had a stroke benefit from opportunities to practice the activities they need to re-learn. It is common practice to give patients written exercises to guide their practice out of therapy session. Whilst more practice is better, it is important that the activities are practiced accurately, to ensure that the right movement patterns are re-learned.

The aim of this study, is to evaluate whether an intervention providing in-patients who have had a stroke an opportunity to use a simple video guide to help them perform their exercises accurately would improve clinical outcomes. Watching an activity being performed helps you to learn the activity more effectively. The focus of this study is arm rehabilitation.

The participants will be adult in-patients in Leeds Teaching Hospitals Trust, and will have had a first time stroke that has left them with some arm weakness.

The participants will be matched according to the severity of their weakness, then randomly allocated to either a treatment as usual group, or an intervention group. Those in the intervention group will have their exercises for their arm and hand recorded onto a tablet during their normal therapy session. They will then be lent the tablet for the duration of the trial, so they can have a visual guide to help them throughout the trial period. Ward staff will be shown how to use the tablet to help any participants who struggle with the technology.

Measurements will be made before and after the trial period to look at ability to move the arm and hand, quality of movement, self-efficacy and time spent exercising. Participants and staff will be asked for their experiences of the intervention or normal practice.

This is a feasibility study with an embedded process evaluation.

DETAILED DESCRIPTION:
This is a small single blind RCT. The outcome assessor will be blinded to the participants status as either in the treatment as usual group or the intervention group. As a feasibility study conducted as part of the development, and planned larger evaluation, of a complex intervention we have drawn heavily on the MRC guidance on complex interventions and process evaluation.

All participants will have the capacity to make an informed decision to consent.

The participants who are suitable to be included in the study will be consented by the student researcher (with support from the Speech and language therapist if needed). This will be done in accordance with the process described in section A27-1.

To reduce the possibility of patients who have severe impairment or other excluding factors being approached an initial screening will have occurred by the direct clinical care team of the potential participants medical notes. This occurs as part of their normal initial assessment of the patient.

Eight patients with mild upper limb impairment will be recruited and eight with moderate upper limb impairment. (Three of each category for both treatment as usual and intervention group).

A tally will be kept of those with mild and moderate weakness in their upper limb, and recruitment will cease once eight participants of each category have been consented. The trial period will commence as a rolling start, with each person starting the trial period as soon as their 'matched pair' has been recruited. Each of the matched pair will be randomly allocated into either control or intervention group.

Once the participants have been consented, they will undergo their baseline assessments. This will be carried out by an experienced neurological physiotherapist from another ward (Blinded to the randomisation into the control or intervention group). The assessment session will be carried out in one of the ward rehabilitation rooms, and is predicted to take no more than half an hour, though more time will be allowed should the participant have further questions.

The patients in the control group will then have their therapy programme as normal for the next four weeks, or until discharge, whichever comes sooner.

The patients in the intervention group will have their next therapy session in the normal manner, but during or at the end of the session,(whichever is most appropriate) the exercises prescribed by the therapist will be filmed onto a tablet. It will consist of the therapist performing the exercise three times to allow the participant to get the idea of the correct movement, and then the participant performing the action three times with the therapist giving verbal prompts to correct the movement.For the intervention group the therapist will be asked to film any upper limb exercises prescribed onto an i-pad, which will provided (one for each patient). Filming will be from two to three feet away, and from whatever angle the physiotherapist feels is most appropriate. The video need not include all of the patient or physiotherapist demonstrator, but should include as much of their body as the therapist feels is needed for guidance.

The i-pad can then be taken by the patient to be used by their bedside. Participants will be given a prompt sheet for playing back their exercises, and the I-pad interface will have been developed with The University of Leeds School of Medicine technology department to make it as intuitive as possible.

For both patient groups, if the therapist would normally provide a written exercise sheet this will also be provided.

The exercises prescribed will be updated by the therapist as deemed appropriate according to the participants needs, either by re-recording them in a subsequent session, and/or updating written exercise sheets.

The participants in the intervention group will have access to the tablet they are using for the duration of the study, labelled and kept in their private bedside locker. Ward staff will be prompted to ensure that during the day if a patient wishes to do their exercises they are 'set up' to do so, either by ensuring exercise sheets are to hand, or the tablet is within reach, and if necessary switched on and opened, with prompts how to start the video (as the technology may be unfamiliar to the patients.) Ward staff will also ensure the tablets are regularly charged.

At the end of the four week period, or up to 72 hours before discharge, the baseline assessment barrage will be repeated by the baseline assessor (still blinded, participants prompted not to divulge group allocation) In order to evaluate the experience of exercising out of therapy sessions, the research physiotherapist will conduct a one to one interview with some of the patient participants. They will be selected via purposive sampling, accounting for initial weakness category and previous experience of using tablet technology. Open ended questions will be used to find out how easy they found it to exercise their affected arm out of therapy time.

Questions asked will be:

* What factors made it difficult to exercise out of therapy time?
* How did you cope using the tablet? (intervention group only)
* Did the video guide influence how you performed the exercises?(intervention group only)
* What suggestions do you have to make using the tablet or video guide better?

Therapy staff will be asked in a focus group setting:

* How useful do you think the video guide was in helping your patients carry out practice out of therapy sessions?
* How did filming the exercises impact on their normal therapy sessions?
* Do they think this intervention could work in practice?
* What would need to change to make it work?

Interviews with patient participants will be carried out in the treatment rooms or by the patients bed if this is their preference.

The Physiotherapy team focus group will be carried out in one of the available treatment rooms.

Patient participants will be asked if they wish to have feedback on the study, and if so home or discharge destination contact details will be recorded, and kept securely, so the participants can receive a written summary of the outcome after the student write up.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18 or over with capacity to give informed consent (according to the mental capacity act 2005) Clinically diagnosed with a first time stroke (To reduce the impact of previous training and rehabilitation interventions) (Stroke physician, from medical notes) Hospitalised patient, staying on a stroke rehabilitation ward. Moderate or mild unilateral upper limb paresis, with minimal inattention.(Therapist assessment)(Mild MSS15-29, Moderate MSS scale ≥30 ) Medically stable and physically capable of participating in active rehabilitation (Ward Doctor) Able to understand consent process and communicate such i.e. minimal aphasic symptoms, able to understand English language enough to consent. (Ward therapists with advice from speech and language therapist where appropriate) No previous significant upper limb pathology that may impact on the participants ability to complete activities Discussion with patient and medical notes review) No Hemi-paretic shoulder pain. (Therapist assessment) Signed informed consent to participate in the trial Active rehabilitation goals, and deemed fit and appropriate for rehabilitation by the therapy team.

Exclusion Criteria:

- Second or more stroke (Stroke physician, from medical notes) Likely to be discharged within two weeks of commencement of trial (It is not always apparent how long someone will remain an in-patient and depends not only on disability, but also social circumstances and patient wishes- therapists judgement for this.(MDT assessment) Age below 18 years Unable to give informed consent. Psychiatric or depressive symptoms that may affect the participants ability to consent or complete the intervention activities(ward Dr) Participation in another clinical trial. Significant apraxia making independent exercise practice difficult (Occupational therapist /physiotherapist judgement) Visual impairment impacting on ability to observe video (Ward team)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Motor status score (MSS) | 4 weeks
  Measures shoulder, elbow wrist hand and finger movements.

SECONDARY OUTCOMES:
Leeds Movement performance Index | 4 weeks
  Measures quality of movement
Time | 4 weeks
  Time spent exercising out of therapy
Generalised self efficacy score (GSE) | 4 weeks
  Measures self - efficacy

IPD SHARING:
Plan to Share IPD: No